CLINICAL TRIAL: NCT06767644
Title: the Effect of Music on Pain and Anxiety During Diagnostic Outpatient Hysteroscopy in Postmenopausal Women: a Randomized Controlled Trial
Brief Title: The Effect of Music on Pain and Anxiety During Diagnostic Outpatient Hysteroscopy in Postmenopausal Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MUSIC POSTMENOPAUSE
Record Dates: First submitted 2025-01-04; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Hysteroscopy
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music group (Experimental)
  Interventions: Other: music
- non-music group (Placebo Comparator)
  Interventions: Other: no music

INTERVENTIONS:
Other: music — In the music group, music chosen by the participant will be played through a speaker by the nursing staff during outpatient hysteroscopy. Music will be played through a speaker instead of headphones in order to maintain good communication and interaction between the participant and the doctor.
  Arms: music group
Other: no music — Participants in the non-music group will undergo outpatient hysteroscopy in the same setting and standard procedure without listening to any music.
  Arms: non-music group

SUMMARY:
This study aims to demonstrate the value of music in diagnostic outpatient hysteroscopy on patients' level of pain and anxiety in postmenopausal women

DETAILED DESCRIPTION:
This study aims to demonstrate the value of music in diagnostic outpatient hysteroscopy on patients' levels of pain and anxiety in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal patients with an indication for ofﬁce hysteroscopy (postmenopausal bleeding or abnormal ultrasound ﬁndings)

Exclusion Criteria:

patients with cervical pathology retroverted uterus (detected by transvaginal ultrasound) previous cervical surgery patients with severe vaginal bleeding

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain | 5 minutes
  Pain intensity will be assessed by visual analog scale during the procedure. visual analog scale ranging from 0 to 10

SECONDARY OUTCOMES:
anxiety during procedure | 5 minutes
  anxiety will be measured using 10 cm VAS like score where 0 denotes no anxiety and 10 represents maximum anxiety

IPD SHARING:
Plan to Share IPD: Undecided